CLINICAL TRIAL: NCT04546724
Title: A Multicenter, Randomized, Placebo-Controlled, Double-Blinded Pivotal Study To Evaluate Safety And Immunogenicity Of A Live-Attenuated Chikungunya Virus Vaccine Candidate In Adults Aged 18 Years And Above
Brief Title: Pivotal Study to Evaluate Safety and Immunogenicity of a Live-Attenuated Chikungunya Virus Vaccine Candidate in Adults
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Valneva Austria GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: VLA1553-301
Record Dates: First submitted 2020-09-04; First posted 2020-09-14 (Actual); Results first posted 2022-07-25 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Chikungunya Virus Infection
Keywords: VLA1553; Chikungunya Virus Infection; CHIKV; Live-attenuated Chikungunya virus vaccine
MeSH Terms: conditions — Chikungunya Fever

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- VLA1553 (Active Comparator): Single intramuscular vaccination on Day 1 with VLA1553, a lyophilized live-attenuated Chikungunya vaccine candidate; 1x10E4 TCID50 per dose
  Interventions: Biological: VLA1553
- Placebo (Placebo Comparator): Single intramuscular vaccination on Day 1 with Phosphate-Buffered Saline (PBS) as placebo
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: VLA1553 — Single intramuscular vaccination on Day 1 with VLA1553, a lyophilized live-attenuated Chikungunya vaccine candidate; 1x10E4 TCID50 per dose
  Arms: VLA1553
Biological: Placebo — Single intramuscular vaccination on Day 1 with Phosphate-Buffered Saline (PBS) as placebo
  Arms: Placebo

SUMMARY:
This was a prospective, randomized, double-blinded, multicenter, pivotal clinical study evaluating the final dose of VLA1553 (1 x10E4 TCID50 per dose) in comparison to a placebo control. The final dose of VLA1553 or control was administered as single immunization on Day 1. Overall, 4.128 male and female subjects aged 18 years and above were randomized into the study.

DETAILED DESCRIPTION:
This was a prospective, double-blinded, multicenter, randomized, pivotal Phase 3 study and 4.128 participants aged 18 years or above were randomized in a 3:1 ratio to the live-attenuated CHIKV vaccine candidate (VLA1553) or placebo. The final dose of lyophilized VLA1553 or placebo was administered as a single intramuscular immunization. Subjects in this study were stratified into two age strata of 18 to 64 years and 65 years of age or above. The primary objective of the study was to evaluate the immunogenicity and safety of the final dose of VLA1553 28 days following the single immunization. Immunogenicity evaluations in the immunogenicity subset included the proportion of subjects with seroprotective neutralizing CHIKV antibody titers above a surrogate threshold indicative of protection. The surrogate of protection reasonably likely to predict clinical benefit has been established in non-human primate passive transfer studies using human sera from the Phase 1 study and was supported by sero-epidemiological studies. Safety data collection and immunogenicity were assessed until Month 6.

The first enrolled and randomized 501 subjects comprised the immunogenicity subset.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or above on the Day of screening
2. able to provide informed consent
3. generally healthy as determined by the Investigator's clinical judgement based on medical history, physical examination and screening laboratory tests
4. for women of childbearing potential:

   1. practiced an adequate method of contraception during 30 days before screening
   2. negative serum or urine pregnancy test at screening
   3. agreed to employ adequate birth control measures for the first three months post-vaccination.

Main Exclusion Criteria:

1. CHIKV infection in the past, including suspected CHIKV infection; was taking medication or other treatment for unresolved symptoms attributed to a previous CHIKV infection; or had participated in a clinical study involving an investigational CHIKV vaccine
2. acute or recent infection
3. Subject tested positive for human immunodeficiency virus (HIV), hepatitis B surface antigen (HBsAg) or hepatitis C virus (HCV);
4. live virus vaccine within 28 days or inactivated vaccine within 14 days prior to vaccination in this study or planned to receive a vaccine within 28 days or 14 days after vaccination, respectively
5. abnormal findings in any required study investigations (including medical history, physical examination, and clinical laboratory) considered clinically relevant by the Investigator which pose a risk for participation in the study
6. medical history of or currently had acute or progressive, unstable or uncontrolled clinical conditions that posed a risk for participation in the study
7. history of immune-mediated or clinically relevant arthritis / arthralgia
8. history of malignancy in the past 5 years other than squamous cell or basal cell skin cancer. If there had been surgical excision or treatment more than 5 years ago that was considered to have achieved a cure, the subject could be enrolled.
9. known or suspected defect of the immune system, such as subjects with congenital or acquired immunodeficiency, including infection with HIV, status post organ transplantation or immuno-suppressive therapy within 4 weeks prior to vaccination.
10. history of any vaccine related contraindicating event (e.g., anaphylaxis, allergy to components of the candidate vaccine, other known contraindications)
11. with clinical conditions representing a contraindication to intramuscular vaccination and blood draws
12. pregnant or lactating at the time of enrollment
13. Donation of blood, blood fractions or plasma within 30 days or received blood-derived products (e.g. plasma) within 90 days prior to vaccination in this study or planned to donate blood or used blood products until Day 180 of the study
14. rash, dermatological condition or tattoos that would, in the opinion of the Investigator, interfere with injection site reaction rating
15. known or suspected problem with alcohol or drug abuse as determined by the Investigator
16. any condition that, in the opinion of the Investigator, could compromise the subjects well-being, interfere with evaluation of study endpoints, or would limit the subject's ability to complete the study;
17. committed to an institution (by virtue of an order issued either by the judicial or the administrative authorities)
18. Participation in another clinical study involving an investigational medicinal product (IMP) or device within 30 days prior to study enrollment or is scheduled to participate in another clinical study involving an IMP, or device during the course of this study
19. member of the team conducting the study or in a dependent relationship with one of the study team members. Dependent relationships include close relatives (i.e., children, partner/spouse, siblings, parents) as well as employees of the Investigator or site personnel conducting the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4128 (Actual)
Dates: Start 2020-09-17 (Actual); Primary Completion 2021-05-19 (Actual); Study Completion 2021-10-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Valneva Clinical Development, Study Chair — Valneva Austria GmbH
Locations (44):
- United States (44):
  - Accelerated Enrollment Solutions (AES), Chandler, Arizona
  - Accelerated Enrollment Solutions (AES), Phoenix, Arizona
  - Alliance for Multispecialty Research (AMR), Tempe, Arizona
  - ELITE Research Network (ELITE), Little Rock, Arkansas
  - Velocity Clinical Research, Chula Vista, Chula Vista, California
  - Accelerated Enrollment Solutions (AES), San Diego, California
  - Accel Research Sites - DeLand, DeLand, Florida
  - ELITE Research Network (ELITE), Hallandale, Florida
  - Meridien Research - Maitland, Maitland, Florida
  - Accelerated Enrollment Solutions (AES), Melbourne, Florida
  - Suncoast Research Group, LLC, Miami, Florida
  - ELITE Research Network (ELITE), North Miami Beach, Florida
  - Jacksonville Center for Clinical Research, LTD dba St. Johns Center for Clinical Research, Ponte Vedra, Florida
  - Synexus - The Villages, The Villages, Florida
  - ELITE Research Network (ELITE), Meridian, Idaho
  - Accelerated Enrollment Solutions (AES), Chicago, Illinois
  - Accelerated Enrollment Solutions (AES), Peoria, Illinois
  - Alliance for Multispecialty Research (AMR), El Dorado, Kansas
  - Alliance for Multispecialty Research (AMR), Newton, Kansas
  - Alliance for Multispecialty Research (AMR), Wichita, Kansas
  - Alliance for Multispecialty Research (AMR), Lexington, Kentucky
  - AMR - New Orleans - Center for Clinical Research, New Orleans, Louisiana
  - Alliance for Multispecialty Research (AMR), Kansas City, Missouri
  - Meridian Clinical Research - Grand Island, Grand Island, Nebraska
  - Platinum Research Network (Platinum), Omaha, Nebraska
  - Accelerated Enrollment Solutions (AES), Omaha, Nebraska
  - Alliance for Multispecialty Research (AMR), Las Vegas, Nevada
  - Meridian Clinical Research, Endwell, New York
  - Rochester Clinical Research, Rochester, New York
  - Lucas Research, Morehead City, North Carolina
  - ELITE Research Network (ELITE), Wilmington, North Carolina
  - Accelerated Enrollment Solutions (AES), Cincinnati, Ohio
  - ELITE Research Network (ELITE), Oklahoma City, Oklahoma
  - Velocity Clinical Research - Medford, Medford, Oregon
  - Synexus - Anderson, Anderson, South Carolina
  - Vitalink Research - Anderson, Anderson, South Carolina
  - Alliance for Multispecialty Research (AMR), Knoxville, Tennessee
  - Tekton Research - Beaumont, Beaumont, Texas
  - PanAmerican Clinical Research - US Headquarter, Brownsville, Texas
  - Velocity Clinical Research - Austin, Cedar Park, Texas
  - Research Your Health, LLC, Plano, Texas
  - ELITE Research Network (ELITE), Tomball, Texas
  - ELITE Research Network (ELITE), West Jordan, Utah
  - Alliance for Multispecialty Research (AMR), Norfolk, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kosulin K, Brasel TL, Smith J, Torres M, Bitzer A, Dubischar K, Buerger V, Mader R, Weaver SC, Beasley DWC, Hochreiter R. Cross-neutralizing activity of the chikungunya vaccine VLA1553 against three prevalent chikungunya lineages. Emerg Microbes Infect. 2025 Dec;14(1):2469653. doi: 10.1080/22221751.2025.2469653. Epub 2025 Mar 10. PMID 39998495
- [Derived] Schneider M, Narciso-Abraham M, Hadl S, McMahon R, Toepfer S, Fuchs U, Hochreiter R, Bitzer A, Kosulin K, Larcher-Senn J, Mader R, Dubischar K, Zoihsl O, Jaramillo JC, Eder-Lingelbach S, Buerger V, Wressnigg N. Safety and immunogenicity of a single-shot live-attenuated chikungunya vaccine: a double-blind, multicentre, randomised, placebo-controlled, phase 3 trial. Lancet. 2023 Jun 24;401(10394):2138-2147. doi: 10.1016/S0140-6736(23)00641-4. Epub 2023 Jun 12. PMID 37321235

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | VLA1553 | Placebo
Started (In total, 4,128 subjects were randomized, of whom 3,093 subjects were randomized in the VLA1553 arm and 1,035 subjects in the placebo arm. Ten subjects in VLA1553 arm and 1 in placebo arm did not receive their vaccination. All vaccinated subjects were included in the Safety population, except for 1 subject that was vaccinated twice.) | 3082 | 1033
Completed | 2724 | 920
Not Completed | 358 | 113
Not completed — Withdrawal by Subject | 145 | 41
Not completed — Adverse Event | 1 | 1
Not completed — Lost to Follow-up | 186 | 63
Not completed — Physician Decision | 8 | 2
Not completed — Death | 2 | 1
Not completed — subject has been out of town | 1 | 0
Not completed — subject is incarcerated | 2 | 0
Not completed — subject is relocating | 12 | 4
Not completed — Subject in another study | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | VLA1553 | Placebo | Total
Number analyzed (Participants) | 3082 | 1033 | 4115
Age, Continuous [Mean (Standard Deviation); unit: years] | 45.1 (15.44) | 45.0 (15.59) | 45.0 (15.47)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1682 | 569 | 2251
  Male | 1400 | 464 | 1864
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 27 | 5 | 32
  Asian | 51 | 17 | 68
  Black or African American | 451 | 122 | 573
  Native Hawaiian or other Pacific Islander | 13 | 5 | 18
  White | 2456 | 853 | 3309
  Other | 84 | 31 | 115

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Seroprotective CHIKV Antibody Level for Baseline Negative Subjects 28 Days Post-vaccination
Description: Seroprotection rate, based on a surrogate of protection agreed with FDA
  Assay used for analysis was based on µPRNT (Micro Plaque Reduction Neutralization Test). Participants at pre-selected sites were included, if they had available Day 1 and Day 29 samples and without major protocol deviations that could impact the immune response.
Time Frame: on Day 29 after single vaccination
Population: The Per-Protocol population used for immunogenicity analyses, is based on participants without major protocol deviations that could impact the immune response.
Measure: Count of Participants; unit: Participants
Groups:
- VLA1553 18-64 Years; VLA1553 ≥65 Years: VLA1553: Single intramuscular vaccination on Day 1 with VLA1553, a lyophilized live-attenuated Chikungunya vaccine candidate; 1x10E4 TCID50 per dose
- Placebo 18-64 Years; Placebo ≥65 Years: Placebo: Single intramuscular vaccination on Day 1 with Phosphate-Buffered Saline (PBS) as placebo
Arm/Group | VLA1553 18-64 Years | Placebo 18-64 Years | VLA1553 ≥65 Years | Placebo ≥65 Years
Number analyzed (Participants) | 207 | 73 | 59 | 23
Participants | 204 | 0 | 59 | 0

2. Secondary Outcome: CHIKV-specific Neutralizing Antibody Titers
Description: CHIKV-specific Neutralizing Antibody Titers on Day 8, and Day 29 Postvaccination as Determined by μPRNT ( (Micro Plaque Reduction Neutralization Test) Assay
Time Frame: Until Day 180
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: Antibody Titers
Arm/Group | VLA1553 18-64 Years | Placebo 18-64 Years | VLA1553 ≥65 Years | Placebo ≥65 Years
Number analyzed (Participants) | 207 | 73 | 59 | 23
Antibody Titers
  Visit 2 - Day 8 | 13.6 [12.22 to 15.23] | 10.2 [9.92 to 10.50] | 13.4 [11.05 to 16.31] | 10.0 [10.0 to 10.0]
  Visit 3 - Day 29 | 3273.7 [2860.93 to 3746.04] | 10.1 [9.89 to 10.33] | 3688.8 [2938.94 to 4630.10] | 10.0 [10.0 to 10.0]
  Visit 4 - Day 85 | 1068.7 [934.77 to 1221.82] | 10.0 [10.0 to 10.0] | 1140.9 [942.97 to 1380.31] | 10.7 [9.71 to 11.78]
  Visit 5 - Day 180 | 755.1 [656.01 to 869.16] | 10.0 [10.0 to 10.0] | 742.8 [578.36 to 954.0] | 10.0 [10.0 to 10.0]

3. Secondary Outcome: Number of Participants With Seroprotective CHIKV Antibody Level
Description: Seroprotection rate, based on a surrogate of protection agreed with FDA Seroprotective CHIKV Antibody Level Defined as μPRNT (Micro Plaque Reduction Neutralization Test) for Baseline Negative Subjects
Time Frame: Until Day 180
Population: The Per-Protocol population used for immunogenicity analyses, is based on participants without major protocol deviations (PDs) that could impact the immune response.
  Counts of participants per time point vary: baseline AND post-line µPRNT result are needed at a given timepoint; results for a specific timepoint were excluded in case of major PD (e.g., major time window deviation resulted in exclusion of a result for a given visit/ time point, results from earlier/ later visits were included)
Measure: Count of Participants; unit: Participants
Arm/Group | VLA1553 18-64 Years | Placebo 18-64 Years | VLA1553 ≥65 Years | Placebo ≥65 Years
Number analyzed (Participants) | 207 | 73 | 59 | 23
Participants
  Visit 2 - Day 8: number analyzed (Participants) | 198 | 70 | 53 | 23
  Visit 2 - Day 8 | 2 | 0 | 2 | 0
  Visit 4 - Day 85: number analyzed (Participants) | 194 | 69 | 52 | 22
  Visit 4 - Day 85 | 189 | 0 | 52 | 0
  Visit 5 - Day 180: number analyzed (Participants) | 184 | 68 | 58 | 23
  Visit 5 - Day 180 | 178 | 0 | 55 | 0

4. Secondary Outcome: Number of Participants With Seroconversion
Description: Seroconversion was defined as CHIKV-specific neutralizing antibody titer of ≥ 20 based on µPRNT (Micro Plaque Reduction Neutralization Test) for baseline negative subjects
Time Frame: Until Day 180
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | VLA1553 18-64 Years | Placebo 18-64 Years | VLA1553 ≥65 Years | Placebo ≥65 Years
Number analyzed (Participants) | 207 | 73 | 59 | 23
Participants
  Visit 3 - Day 29 | 205 | 1 | 59 | 0
  Visit 5 - Day 180: number analyzed (Participants) | 184 | 68 | 58 | 23
  Visit 5 - Day 180 | 181 | 0 | 57 | 0

5. Secondary Outcome: Fold "Change" of CHIKV-specific Neutralizing Antibody Titers Compared to Baseline
Description: Fold Change of CHIKV-specific Neutralizing Antibody Titers Determined by μPRNT ( (Micro Plaque Reduction Neutralization Test) as compared to baseline
Time Frame: until Day 180
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: fold increase
Arm/Group | VLA1553 18-64 Years | Placebo 18-64 Years | VLA1553 ≥65 Years | Placebo ≥65 Years
Number analyzed (Participants) | 207 | 73 | 59 | 23
fold increase
  Visit 3 - Day 29 | 460.27 (384.052) | 1.02 (0.140) | 507.70 (412.467) | 1.00 (0.000)
  Visit 5 - Day 180: number analyzed (Participants) | 184 | 68 | 58 | 23
  Visit 5 - Day 180 | 108.81 (97.238) | 1.00 (0.000) | 102.09 (79.433) | 1.00 (0.000)

6. Secondary Outcome: Number of Participants Reaching an X-fold Change in CHICKV-specific Neutralizing Antibody Titer Compared to Baseline
Description: Number of Participants Reaching an at Least 4-fold, 8-fold, 16-fold or 64-fold change of CHIKV-specific Neutralizing Antibody Titers Determined by μPRNT ( (Micro Plaque Reduction Neutralization Test) as compared to baseline
Time Frame: until Day 180
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | VLA1553 18-64 Years | Placebo 18-64 Years | VLA1553 ≥65 Years | Placebo ≥65 Years
Number analyzed (Participants) | 207 | 73 | 59 | 23
Participants
  Visit 3 - Day 29: Subjects reaching 4-fold increase | 205 | 0 | 59 | 0
  Visit 3 - Day 29: Subjects reaching 8-fold increase | 205 | 0 | 59 | 0
  Visit 3 - Day 29: Subjects reaching 16-fold increase | 204 | 0 | 59 | 0
  Visit 3 - Day 29: Subjects reaching 64-fold increase | 200 | 0 | 57 | 0
  Visit 5 - Day 180: Subjects reaching 4-fold increase: number analyzed (Participants) | 184 | 68 | 58 | 23
  Visit 5 - Day 180: Subjects reaching 4-fold increase | 181 | 0 | 57 | 0
  Visit 5 - Day 180: Subjects reaching 8-fold increase: number analyzed (Participants) | 184 | 68 | 58 | 23
  Visit 5 - Day 180: Subjects reaching 8-fold increase | 181 | 0 | 56 | 0
  Visit 5 - Day 180: Subjects reaching 16-fold increase: number analyzed (Participants) | 184 | 68 | 58 | 23
  Visit 5 - Day 180: Subjects reaching 16-fold increase | 177 | 0 | 55 | 0
  Visit 5 - Day 180: Subjects reaching 64-fold increase: number analyzed (Participants) | 184 | 68 | 58 | 23
  Visit 5 - Day 180: Subjects reaching 64-fold increase | 106 | 0 | 35 | 0

7. Secondary Outcome: Unsolicited AEs
Description: Number of Participants with Unsolicited Adverse Events
Time Frame: Until Day 29
Measure: Count of Participants; unit: Participants
Arm/Group | VLA1553 | Placebo
Number analyzed (Participants) | 3082 | 1033
Participants | 687 | 138

8. Secondary Outcome: Solicited Injection Site AEs
Description: Number of Participants with solicited injection site reactions
Time Frame: within 10 days post-vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | VLA1553 | Placebo
Number analyzed (Participants) | 3082 | 1033
Participants
  Any Solicited Injection Site Adverse Event | 463 | 115
  Tenderness | 328 | 84
  Pain | 191 | 38
  Erythema/Redness | 46 | 15
  Induration | 44 | 8
  Swelling | 21 | 8

9. Secondary Outcome: Solicited Systemic AEs
Description: Number of Participants with solicited systemic reactions
Time Frame: within 10 days post-vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | VLA1553 | Placebo
Number analyzed (Participants) | 3082 | 1033
Participants
  Any Solicited Systemic Adverse Event | 1547 | 278
  Headache | 969 | 151
  Fatigue | 879 | 130
  Myalgia | 735 | 76
  Arthralgia | 520 | 50
  Fever | 414 | 8
  Nausea | 345 | 58
  Rash | 70 | 5
  Vomiting | 58 | 10

10. Secondary Outcome: Adverse Events
Description: Number of Participants with any Adverse Events
Time Frame: until Day 180
Measure: Count of Participants; unit: Participants
Arm/Group | VLA1553 | Placebo
Number analyzed (Participants) | 3082 | 1033
Participants
  Mild | 1287 | 336
  Moderate | 532 | 112
  Severe | 104 | 14

11. Secondary Outcome: Related Adverse Events
Description: Number of Participants with any related Adverse Events
Time Frame: until Day 180
Measure: Count of Participants; unit: Participants
Arm/Group | VLA1553 | Placebo
Number analyzed (Participants) | 3082 | 1033
Participants | 1575 | 322

12. Secondary Outcome: Serious Adverse Event
Description: Number of Participants with any Serious Adverse Events
Time Frame: until Day 180
Measure: Count of Participants; unit: Participants
Arm/Group | VLA1553 | Placebo
Number analyzed (Participants) | 3082 | 1033
Participants | 46 | 8

13. Secondary Outcome: Related Serious Adverse Event
Description: Number of Participants with any Related Serious Adverse Events
Time Frame: until Day 180
Measure: Count of Participants; unit: Participants
Arm/Group | VLA1553 | Placebo
Number analyzed (Participants) | 3082 | 1033
Participants | 2 | 0

14. Secondary Outcome: Adverse Event of Special Interest
Description: Number of Participants with any Adverse Event of Special Interest
  AESI Definition:
  The following cluster of symptoms suggestive of CHIKV infection with or without remissions or exacerbations received particular consideration:
  1. Fever (≥38.0°C [100.4°F] measured orally) and
  2. Acute (poly)arthralgia/arthritis most frequently in the extremities (wrists, ankles, and phalanges, often symmetric), back pain and/or neurological symptoms (e.g. confusion, optic neuritis, meningoencephalitis, or polyneuropathy) and/or cardiac symptoms (e.g. myocarditis) or One or more of the following signs and symptoms: macular to maculopapular rash (sometimes with cutaneous pruritus [foot plant] and edema of the face and extremities), polyadenopathies; and
  3. Onset of symptoms 2 to 21 days after vaccination and
  4. Duration of event ≥3 days.
Time Frame: within 21 days post-vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | VLA1553 | Placebo
Number analyzed (Participants) | 3082 | 1033
Participants | 10 | 1

15. Secondary Outcome: Related Adverse Event of Special Interest
Description: Number of Participants with any Related Adverse Event of Special Interest
  AESI Definition:
  The following cluster of symptoms suggestive of CHIKV infection with or without remissions or exacerbations received particular consideration:
  1. Fever (≥38.0°C [100.4°F] measured orally) and
  2. Acute (poly)arthralgia/arthritis most frequently in the extremities (wrists, ankles, and phalanges, often symmetric), back pain and/or neurological symptoms (e.g. confusion, optic neuritis, meningoencephalitis, or polyneuropathy) and/or cardiac symptoms (e.g. myocarditis) or One or more of the following signs and symptoms: macular to maculopapular rash (sometimes with cutaneous pruritus [foot plant] and edema of the face and extremities), polyadenopathies; and
  3. Onset of symptoms 2 to 21 days after vaccination and
  4. Duration of event ≥3 days.
Time Frame: within 21 days post-vaccination
Measure: Count of Participants; unit: Participants
Arm/Group | VLA1553 | Placebo
Number analyzed (Participants) | 3082 | 1033
Participants | 9 | 1

ADVERSE EVENTS:
Time Frame: Day 180
Description: Solicited AEs are collected by systematic assessment through subject eDiaries (within 10 days post-vaccination):injection site AEs (pain, tenderness, induration, swelling, erythema/redness) or systemic AEs (headache, myalgia, arthralgia, fever, vomiting, nausea, rash, fatigue). Unsolicited AEs, and SAEs are collected by non-systematic assessment up to Day 180.
  AESI is defined as symptoms suggestive of CHIKV infection up to 21 days after vaccination and collected by systematic assessment.
Arm/Group | VLA1553 | Placebo
All-Cause Mortality (participants affected / at risk) | 2/3082 | 1/1033
Serious Adverse Events (participants affected / at risk) | 46/3082 | 8/1033
Other Adverse Events (participants affected / at risk) | 1721/3082 | 373/1033
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VLA1553 (N=3082) | Placebo (N=1033)
Appendicitis (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 (Infections and infestations) | 1 (1) | 1 (1)
Complicated appendicitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia (Infections and infestations) | 2 (2) | 1 (1)
Pyelonephritis (Infections and infestations) | 1 (1) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ankle fracture (Injury, poisoning and procedural complications) | 2 (3) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Tibia fracture (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 3 (3) | 1 (1)
Anxiety (Psychiatric disorders) | 0 (0) | 1 (2)
Depression (Psychiatric disorders) | 3 (3) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 1 (1) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 1 (1) | 0 (0)
Hydronephrosis (Renal and urinary disorders) | 1 (1) | 0 (0)
Nephrolithiasis (Renal and urinary disorders) | 1 (1) | 0 (0)
Atrial fibrillation (Cardiac disorders) | 2 (4) | 0 (0)
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1 (1) | 0 (0)
Gastrointestinal haemorrage (Gastrointestinal disorders) | 0 (0) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1) | 0 (0)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Cerebellar haemorrhage (Nervous system disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)
Arthritis bacterial (Infections and infestations) | 1 (1) | 0 (0)
COVID-19 pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (1) | 0 (0)
Kidney infection (Infections and infestations) | 0 (0) | 1 (1)
Road traffic accident (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haematoma (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Procedural pain (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Splenic rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Traumatic liver injury (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Anxiety disorder (Psychiatric disorders) | 1 (1) | 0 (0)
Depression suicidal (Psychiatric disorders) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 1 (1)
Cardiac arrest (Cardiac disorders) | 1 (1) | 0 (0)
Cardiomyopathy (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 0 (0)
Guillain-Barre syndrome (Nervous system disorders) | 1 (1) | 0 (0)
Neuropathy peripheral (Nervous system disorders) | 1 (1) | 0 (0)
Syncope (Nervous system disorders) | 1 (1) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cannabinoid hyperemesis syndrome (Gastrointestinal disorders) | 1 (1) | 0 (0)
Colitis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 1 (1) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0)
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Non-small cell lung cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0)
Foetal death (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Lumber spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Non-cardiac chest pain (General disorders) | 1 (1) | 0 (0)
Anaphylactic reaction (Immune system disorders) | 1 (1) | 0 (0)
SARS-CoV-2 test positive (Investigations) | 1 (1) | 0 (0)
Prostatomegaly (Reproductive system and breast disorders) | 1 (1) | 0 (0)
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Hypotension (Vascular disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | VLA1553 (N=3082) | Placebo (N=1033)
Headache (Nervous system disorders) | 986 (1028) | 160 (178)
Fatigue (General disorders) | 886 (893) | 137 (139)
Myalgia (Musculoskeletal and connective tissue disorders) | 750 (758) | 82 (84)
Arthralgia (Musculoskeletal and connective tissue disorders) | 554 (589) | 63 (70)
Injection site pain (General disorders) | 413 (519) | 101 (122)
Pyrexia (General disorders) | 427 (429) | 13 (13)
Nausea (Gastrointestinal disorders) | 359 (364) | 63 (64)
Rash (Skin and subcutaneous tissue disorders) | 82 (86) | 12 (12)
COVID-19 (Infections and infestations) | 59 (70) | 22 (23)
Vomiting (Gastrointestinal disorders) | 66 (67) | 14 (14)
Chills (General disorders) | 59 (60) | 3 (3)
Injection site erythema (General disorders) | 47 (47) | 15 (15)
Injection site induration (General disorders) | 44 (44) | 8 (8)
Back pain (Musculoskeletal and connective tissue disorders) | 44 (46) | 7 (7)
Diarrhoea (Gastrointestinal disorders) | 46 (46) | 4 (4)
Urinary tract infection (Renal and urinary disorders) | 33 (36) | 6 (6)
Neutropenia (Blood and lymphatic system disorders) | 34 (34) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-03-23): https://cdn.clinicaltrials.gov/large-docs/24/NCT04546724/Prot_000.pdf
  • Statistical Analysis Plan (2022-01-14): https://cdn.clinicaltrials.gov/large-docs/24/NCT04546724/SAP_001.pdf